CLINICAL TRIAL: NCT05194709
Title: Clinical Trial of Anti-5T4 Oncofetal Trophoblast Glycoprotein (5T4) Conjugated Antibody Redirecting Natural Killer (CAR-NK) Cells in Advanced Solid Tumors
Brief Title: Study of Anti-5T4 CAR-NK Cell Therapy in Advanced Solid Tumors
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wuxi People's Hospital (Other)
Collaborators: Imbioray (Hangzhou) Biomedicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IBR854-T01; WX-IBR-8 (Other: Wuxi People's Hospital)
Record Dates: First submitted 2022-01-04; First posted 2022-01-18 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anti-5T4 CAR-NK Cells (Experimental)
  Interventions: Biological: Anti-CAR-NK Cells

INTERVENTIONS:
Biological: Anti-CAR-NK Cells — The administration of CAR-NK cell will be performed on day 1 and day 3 of each cycle (21 days). The first administration dose in the first cycle is 3.0×10^9 cells. If no adverse events were observed, the second administration dose in the first cycle would be 4.0×10^9 cells, and each administration dose in the second cycle and thereafter would be 4.0×10^9 cells.

SUMMARY:
This study is an interventional, single arm, open-label, investigator-initiated trial (IIT) to evaluate the safety, tolerability, initial efficacy and pharmacokinetics (PK) of anti-5T4 CAR-NK cells in patients with advanced solid tumors.

DETAILED DESCRIPTION:
The treatment cycle in this study is 21 days. The administration of CAR-NK cell will be performed on day 1 and day 3 of each cycle. Subjects will be treated continuously until the criteria for termination of treatment are met. In this study, the dose escalation design is adopted. The first administration dose in the first cycle is 3.0×10^9 cells. If no adverse events were observed, the second administration dose in the first cycle would be 4.0×10^9 cells, and each administration dose in the second cycle and thereafter would be 4.0×10^9 cells.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects volunteer to participate in this clinical study, are fully aware of the study and have signed the Informed Consent Form (ICF). Subjects are willing to follow and able to complete all trial procedures.
2. Age: adult at the age of 18-80 (both inclusive), female or male.
3. Patients with advanced malignant solid tumors, histologically or cytologically confirmed, who had failed standard therapy, or had no standard therapy, or were not eligible for standard therapy at this stage; tumor biomarkers combined with imaging can be used to diagnose some special advanced tumors.
4. Eastern Cooperative Oncology Group (ECOG) score ≤2 and expected survival time >3 months.
5. Organ function during screening should meet the following criteria:

   * Absolute neutrophil count (ANC)≥0.8×109/L
   * Platelet (PLT)≥50×109/L
   * Hemoglobin (Hb)≥80g/L
   * Total bilirubin (TBIL)≤2×ULN
   * Alanine aminotransferase (ALT)≤3×ULN; Patients with liver metastasis or liver cancer: ≤5×ULN
   * Aspartate aminotransferase (AST)≤3×ULN; Patients with liver metastasis or liver cancer: ≤5×ULN
   * Creatinine (Cr)≤1.5× ULN
   * Creatinine clearance (Ccr) (to be calculated only when Cr > 1.5× ULN)>50ml/min/1.73m2 (Cockcroft-Gault formula)
   * Activated partial thrombin time (APTT)≤1.5×ULN
   * International normalized ratio (INR)≤1.5×ULN
6. Subjects of reproductive age and their partners should agree to have no family planning and to use effective contraceptive methods (hormonal or barrier methods or abstinence, etc.) for 6 months from signing the ICF until the last dose of the study drug is administered; women of reproductive age should not be pregnant or breastfeeding.

Exclusion Criteria:

1. Have received systemic antitumor therapy, including chemotherapy, immunotherapy, and radical radiotherapy, within 1 week prior to their first use of the study drug.
2. Have participated in other clinical trials and received any unmarketed investigational drug or treatment within 4 weeks prior to first use of the study drug.
3. Any prior adoptive cellular immunotherapy.
4. Have undergone major organ surgery (excluding needle biopsy or surgery related to this indication) within 4 weeks prior to their first use of the study drug, or required elective surgery during the study period.
5. Patients with severe infections that cannot be controlled.
6. Patients with a known history of human immunodeficiency virus (HIV) infection, or a history of organ transplantation.
7. Have active autoimmune diseases or have had autoimmune diseases that are likely to recur (e.g., systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, autoimmune thyroid disease, vasculitis, psoriasis, etc.). Except in the following cases: type 1 diabetes that was well controlled with hormone replacement therapy, hypothyroidism, skin conditions that did not require systemic therapy (e.g., vitiligo), and other conditions that were well controlled and that the investigator determined were less likely to recur (e.g., childhood asthma in remission).
8. Have a history of serious cardiovascular and cerebrovascular diseases, including but not limited to:

   * There are serious cardiac rhythm or conduction abnormalities, such as ventricular arrhythmia, and Ⅱ-Ⅲ degree atrioventricular block, which need clinical intervention;
   * The mean QT interval corrected by Fridericia method (QTcF) is prolonged (male>450ms, female>470ms);
   * Acute coronary syndrome, congestive heart failure, aortic dissection, stroke, or other grade 3 or above cardiovascular and cerebrovascular events occurring within 6 months before the first administration;
   * Patients with heart failure or left ventricular ejection fraction (LVEF) < 50% in the New York Heart Association (NYHA) classification ≥II;
   * Hypertension beyond clinical control.
9. Adverse effects of previous antineoplastic therapy have not returned to CTCAE grade 5.0≤2 (except for toxicity that the investigator determined to be of no safety risk, such as alopecia, hypothyroidism stabilized by hormone replacement therapy).
10. Central nervous system metastases with clinical symptoms.
11. Had other malignant tumors in the past 3 years, excluding skin basal cell carcinoma, ductal carcinoma in situ and cervical carcinoma in situ with a radical surgery.
12. Have a history of alcohol or drug abuse or mental disorder.
13. The investigator considered that the subjects had a history of other serious systemic diseases or other reasons that made them unsuitable for the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-12-30 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse Events (AEs) | From day 1 to day 90 after the last dose
  To evaluate the safety and tolerability of anti-5T4 CAR-NK cells

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 1 year after infusion
  To determine the anti-tumor effectivity of anti-5T4 CAR-NK cells
Progression-free survival (PFS) | Up to 1 year after infusion
  To determine the anti-tumor effectivity of anti-5T4 CAR-NK cells
Overall survival (OS) | Up to 1 year after infusion
  To determine the anti-tumor effectivity of anti-5T4 CAR-NK cells
Disease control rate (DCR) | Up to 1 year after infusion
  To determine the anti-tumor effectivity of anti-5T4 CAR-NK cells
Cytokine release | Up to 1 year
  Blood samples will be collected at specified time points to detect the cytokine (IL-1β, IL-2, IL-4, IL-6, IL-10, IFN-γ, hsCRP) concentration (pg/mL)
Lymphocyte subtype | Up to 1 year
  Blood samples will be collected at specified time points to analyze the lymphocyte subtypes (CD3, CD4, CD8, CD19, CD56)

CONTACTS AND LOCATIONS:
Overall Officials: Peihua P Lu, MD, Principal Investigator — Wuxi People's Hospital
Locations (1):
- Wuxi People's Hospital, Wuxi, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No